CLINICAL TRIAL: NCT01101048
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 167 in Healthy Men and Postmenopausal Women With Low Bone Mineral Density
Brief Title: An Ascending Multiple Dose Study Evaluating AMG 167 in Healthy Men and Postmenopausal Women With Low Bone Mineral Density
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20080389
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Osteopenia
Keywords: Amgen; Phase 1b; Postmenopausal; Bone Mineral Density
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): Two (2) women in each of cohorts 1 and 4, and two (2) men in cohort 2 will receive placebo every 2 weeks for a total of 6 doses. Two (2) women in each of cohorts 3 and 5, and two (2) men in cohort 6 will receive placebo every 4 weeks for a total of 3 doses. Six (6) women in cohort 7 will receive placebo every 2 weeks for a total of 12 doses. In addition, subjects in cohorts 4 have the option to receive an additional 6 doses of placebo; subjects in cohorts 5 and 6 have the option to receive an additional 3 doses. Subjects in cohort 7 have the option to transition to 6 months of alendronate treatment.
  Interventions: Drug: AMG 167
- B (Active Comparator): Six (6) women in each of cohorts 1 and 4, and six (6) men in cohort 2 will receive AMG 167 every 2 weeks for a total of 6 doses. Six (6) women in each of cohorts 3 and 5, and six (6) men in cohort 6 will receive AMG 167 every 4 weeks for a total of 3 doses. Eighteen (18) women in cohort 7 will receive AMG 167 every 2 weeks for a total of 12 doses. In addition, subjects in cohorts 4 have the option to receive an additional 6 doses of AMG 167; subjects in cohorts 5 and 6 have the option to receive an additional 3 doses. Subjects in cohort 7 have the option to transition to 6 months of alendronate treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Subjects will be randomized to receive one of 3 doses of AMG 167 or equivalent volume of placebo administered at once every two-week or once every four-week dosing intervals. Postmenopausal women will receive AMG 167 in one of 3 fixed doses, while men will receive AMG 167 in one of 2 fixed doses by injection under the skin.
  Arms: B
Drug: AMG 167 — Subjects will be randomized to receive one of 3 doses of AMG 167 or equivalent volume of placebo administered at once every two-week or once every four-week dosing intervals. Postmenopausal women will receive AMG 167 in one of 3 fixed doses, while men will receive AMG 167 in one of 2 fixed doses by injection under the skin.
  Arms: A

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and potential immune response of AMG 167 following multiple subcutaneous (SC, injection under the skin) dose administrations in healthy men and postmenopausal women with low bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* Low bone mineral density as determined at the time of screening [as defined by bone mineral density (BMD) T-scores of the lumbar spine (L1-L4), or total evaluable vertebrae (if fewer than L1-L4); or femoral neck between -1.0 and -2.5, exclusive]
* 25-hydroxyvitamin D ≥ 20 ng/mL
* Willing and able to take ≥ 1,000 mg elemental calcium and ≥ 800 IU (but ≤ 1,000 IU) vitamin D daily upon enrollment

Exclusion Criteria:

* Osteoporosis, as defined by BMD T-scores of the lumbar spine (L1-L4) or total evaluable vertebrae (if fewer than L1-L4); or femoral neck ≤ 2.5
* History of vertebral fracture, or fragility fracture (a fracture resulting from no or minor trauma; ie, fall from standing height or less) of the wrist, humerus, hip, or pelvis after age 50
* Diagnosed with any condition that will affect bone metabolism
* Diagnosis of clotting factor deficiency or history of bleeding or coagulation disorder
* History of spinal stenosis
* History of facial nerve paralysis

Exclusion Criteria for Cohort 7 Sub-study (Transition to Alendronate):

* Contraindicated or intolerant of alendronate therapy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The number (percent) of subjects experiencing clinically significant changes in safety laboratory tests, physical examinations, vital signs, or electrocardiograms (ECGs) | 168, 252, or 336 days following initial investigational product administration
The number (percent) of subjects reporting treatment-emergent adverse events | 168, 252, or 336 days following initial investigational product administration
The number (percent) of subjects who develop anti-AMG 167 antibodies | 168, 252, or 336 days following initial investigational product administration

SECONDARY OUTCOMES:
Pharmacodynamic parameters [bone mineral density as assessed by dual energy X-ray absorptiometry (DXA), serum procollagen type 1 N-terminal propeptide (P1NP), osteocalcin, bone-specific alkaline phosphatase (BSAP), and serum CTX levels] and sclerostin | 168, 252, or 336 days following initial investigational product administration
Pharmacokinetics | 168, 252, or 336 days following initial investigational product administration

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com